CLINICAL TRIAL: NCT05981885
Title: 68Ga-FAPI PET/CT to Detect Ongoing Fibroblast Activity in Post-acute COVID-19 With Respiratory Impairment After Hospital Discharge
Brief Title: 68Ga-FAPI PET/CT to Detect Ongoing Fibroblast Activity in Post-acute COVID-19
Acronym: FAPI CLIMATE
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 202100802
Record Dates: First submitted 2023-06-22; First posted 2023-08-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Post-Acute COVID-19; Post-Acute COVID-19 Infection; Post-Acute COVID-19 Syndrome; Pulmonary Fibrosis
Keywords: 68Ga-FAPI-04; HRCT; Post-ICU; Post high-flow Nasal Oxygen therapy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Biospecimen Retention: Samples With DNA — Blood and nose epithelium for single cell RNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the role fibroblasts play in the persistent respiratory complaints after a COVID-19 infection. Fibroblasts are involved in tissue remodeling and repair by creating scar-tissue (fibrosis) after tissue damage has occurred. The hypothesis is that this process of fibrosis is ongoing in patients with persistent complaints. To evaluate the roll of fibroblasts a new type of scan is used that is capable of imaging active fibroblasts, a 68Ga-FAPI PET/CT scan.

DETAILED DESCRIPTION:
Rationale: The pathogenesis of post-acute COVID-19 with respiratory complaints remains unknown. We aim to explore the pulmonary pattern and fibrosis activity in patients with post-acute COVID-19 with respiratory complaints using 68Ga-FAPI Positron Emission Tomography-Computed Tomography (PET/CT) imaging.

Objective: To relate pulmonary fibroblast activity, measured by FAPI-PET/CT at least 3 months after hospital discharge, to interstitial lung abnormalities on high resolution CT (HRCT) at the same time point in post-acute COVID-19 patients with respiratory complaints.

Study design: This is a ZonMw funded single center prospective observational cohort study of post-acute COVID-19 patients with respiratory complaints.

Study population: We will recruit 20 adult patients, all post-ICU or post High-Flow Nasal Oxygen therapy due to there COVID-19 infection, with post-acute COVID-19 and respiratory complaints that will undergo 68Ga-FAPI PET/CT imaging to establish pulmonary fibrosis activity.

Main study parameters/endpoints: To assess the degree of Fibroblast Activation Protein expression on 68Ga-FAPI PET/CT at least 3 months after hospital discharge and to relate this to interstitial lung abnormalities on HRCT at the same time point.

ELIGIBILITY:
Inclusion Criteria:

* Male patients >18 years and female patients >20 years discharged from hospital after PCR-confirmed COVID-19 infection.
* Previous ICU or ward admission with high flow nasal oxygen (HFNO) or mechanical ventilation.
* Persistent respiratory complaints (shortness of breath) at least 3 months after hospital discharge.

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* History of claustrophobia or feeling of inability to tolerate supine position for the PET/CT scans.
* Severe or significant comorbidity, defined as COPD GOLD stage II or higher and/or known interstitial lung disease.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults previously admitted to the ICU or ward requiring mechanical ventilation or high flow nasal oxygen due to their COVID-19 infection with now post-acute COVID-19 and respiratory complaints.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Pulmonary SUV values | At time of inclusion (T0)
  Based on the FAPI PET/CT scan 3-dimensinal volumes of intrest (VOI) are drawn of high FAPI uptake areas (leasions) and non-uptake areas. Using these VOIs SUV values and metabolic active volume (MAV) can be calculated which then can be used to calculate: total lesion FAPI (TL-FAPI), whole-lung FAPI-MAV (wl FAPI-MAV), wlSUVmean and whole lung TL-FAPI (wlTL-FAPI).

SECONDARY OUTCOMES:
Correlate biomarkers to pulmonary SUV values | At time of inclusion (T0)
  A correlation between the pulmonary FAPI uptake, reported as SUV values (see outcome 1) will be correlated with fibrosis and inflammatory specific biomarkers using Pearson's or Spearman's test.
6 minute walking test vs pulmonary SUV values | At time of inclusion (T0)
  The total walked distance in meters during 6 minutes is correlated with pulmonary FAPI uptake, reported as SUV values (see outcome 1) using Pearson's or Spearman's test.
DCLO and VC vs pulmonary SUV values | At time of inclusion (T0)
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated with DCLO and VC using Pearon's or Spearman's test.
Daily impairments (EQ-5D questionnaire) vs pulmonary SUV values | At time of inclusion (T0)
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated with self-reported daily impairments per category as measured by the EQ-5D questionnaire using Pearson's or Spearman's test.
Cellular phenotypes | At time of inclusion (T0)
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated to systemic and upper respiratory tract cellular phenotypes determined by single cell RNA sequencing using Pearon's or Spearmen's test.
HRCT | At time of inclusion (T0)
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated to HRCT findings: extent of disease (0-100%), reticular pattern (0-100%), portion of groundglass (0-100%), coarness (0-3), honey combing (Yes/No), Distribution groundglass, crazy-paving pattern (Yes/No), fibrosis (Yes/No), Bronchiectasis (Yes/No), Emfyseem (Yes/No) and Pleural effusion (Yes/No).
Follow-up HRCT | 10 months after T0
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated to HRCT findings in case of persistent respiratory complaints 8-10 months after T0. Findings that are correlated are: extent of disease (0-100%), reticular pattern (0-100%), portion of groundglass (0-100%), coarness (0-3), honey combing (Yes/No), Distribution groundglass, crazy-paving pattern (Yes/No), fibrosis (Yes/No), Bronchiectasis (Yes/No), Emfyseem (Yes/No) and Pleural effusion (Yes/No).
Follow-up daily impairments (EQ-5D questionnaire) vs pulmonary SUV values | 10 months after T0
  Pulmonary FAPI uptake, reported as SUV values (see outcome 1), will be correlated with self-reported daily impairments per category as measured by the EQ-5D questionnaire using Pearson's or Spearman's test.

CONTACTS AND LOCATIONS:
Overall Officials: Riemer Slart, Prof MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data underlie the results reported in this article will be shared on reasonably request after deidentification of individual participant data. Only investigators whose proposed use of data is for individual participant data meta-analysis and in line with the signed informed consent are eligible for sharing. Proposals should be directed to r.h.j.a.slart@umcg.nl. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Directly after publication
Access Criteria: Only investigators whose proposed use of data is for individual participant data meta-analysis and in line with the signed informed consent are eligible for sharing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05981885/Prot_SAP_000.pdf